CLINICAL TRIAL: NCT00070005
Title: A Phase III Randomised Study Of J-Pouch Coloanal Anastomosis Versus Side-To-End Coloanal Anastomosis After Preoperative Radiotherapy And Total Mesorectal Excision In Patients With Mid And Distal Rectal Cancer
Brief Title: J-Pouch Coloanal Anastomosis Compared With Side-to-End Coloanal Anastomosis After Radiation Therapy and Surgery to Remove the Rectum in Treating Patients With Rectal Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CKTO-2002-02-POCASTER; CDR0000328269 (Registry Identifier: PDQ (Physician Data Query)); EU-20247
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-04

CONDITIONS: Colorectal Cancer; Perioperative/Postoperative Complications
Keywords: perioperative/postoperative complications; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications; Rectal Neoplasms

INTERVENTIONS:
Procedure: conventional surgery
Procedure: management of therapy complications

SUMMARY:
RATIONALE: A coloanal anastomosis may be effective in restoring bowel function after radiation therapy and surgery to remove the rectum. It is not yet known whether a J-pouch coloanal anastomosis is more effective than a side-to-end coloanal anastomosis in restoring bowel function in patients with rectal adenocarcinoma who have undergone radiation therapy and surgery to remove the rectum.

PURPOSE: This randomized phase III trial is studying how well J-pouch coloanal anastomosis works compared to side-to-end coloanal anastomosis in treating patients with rectal adenocarcinoma who have undergone radiation therapy and surgery to remove the rectum.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare functional outcome in patients with mid- or distal rectal adenocarcinoma when treated with J-pouch coloanal anastomosis vs side-to-end coloanal anastomosis after preoperative radiotherapy and total mesorectal excision.

Secondary

* Compare the quality of life of patients treated with these procedures.
* Compare anorectal function in patients treated with these procedures.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and gender. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo total mesorectal excision followed by a J-pouch coloanal anastomosis.
* Arm II: Patients undergo total mesorectal excision followed by a side-to-end coloanal anastomosis.

In both arms, patients receive a temporary ileostomy. The ileostomy is closed after 1 week provided recovery is uneventful and no radiological signs of anastomotic leakage are detected. If early closure is not possible, the ileostomy is closed after 6-8 weeks.

Functional outcome, quality of life, and anorectal function are assessed before surgery and at 4 and 12 months after surgery.

PROJECTED ACCRUAL: A minimum of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * T2 or T3 disease
* Disease located in the mid- or distal rectum
* No evidence of metastatic disease
* No preexisting grade III or IV incontinence
* Completed preoperative radiotherapy (5 x 5 Gy) before study entry

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Working knowledge of the Dutch language

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to the pelvis

Surgery

* No prior colon resection
* No prior anorectal surgery
* No concurrent abdominoperineal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-06

PRIMARY OUTCOMES:
Functional outcome as measured by a validated questionnaire

SECONDARY OUTCOMES:
Quality life as measured by a validated questionnaire
Anorectal function as assessed by anorectal manometry and barostat measurements

CONTACTS AND LOCATIONS:
Overall Officials: Roel Bakx, MD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (9):
- Netherlands (9):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - St. Lucas - Andreas Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Reinier de Graaf Group - Delft, Delft
  - Albert Schweitzerziekenhuis - Locatie Amstelwijck, Dordrecht NM
  - Isala Klinieken - locatie Sophia, Zwolle
  - Isala Klinieken - locatie Weezenlanden, Zwolle